CLINICAL TRIAL: NCT01543204
Title: Open Label Study to Evaluate the Efficacy of Etanercept Treatment in Subjects With Moderate to Severe Plaque Psoriasis Who Have Lost a Satisfactory Response to Adalimumab
Brief Title: Etanercept Treatment in Patients With Moderate to Severe Plaque Psoriasis Who Lost Response to Adalimumab
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision due to slow enrollment
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20101145
Record Dates: First submitted 2012-01-17; First posted 2012-03-02 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Psoriasis
Keywords: plaque psoriasis; etanercept; adalimumab
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept 50 mg (Experimental): Participants received etanercept 50 mg, twice weekly (BIW), subcutaneously (SC) for 12 weeks followed by 50 mg, once weekly (QW), SC for an additional 12 weeks.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Administered by subcutaneous injection
  Other Names: Enbrel®

SUMMARY:
This study will evaluate the efficacy of etanercept in patients with plaque psoriasis who have lost a satisfactory response to adalimumab.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe plaque psoriasis
* Loss of satisfactory response to adalimumab
* Currently receiving or recently discontinued treatment with adalimumab

Exclusion Criteria:

* Active skin conditions that would interfere with evaluations of the effect of investigational product on psoriasis
* Serious medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2015-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (46):
- United States (41):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Encino, California
  - Research Site, Irvine, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, San Ramon, California
  - Research Site, Santa Monica, California
  - Research Site, Denver, Colorado
  - Research Site, Farmington, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Skokie, Illinois
  - Research Site, New Albany, Indiana
  - Research Site, Plainfield, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, East Windsor, New Jersey
  - Research Site, Verona, New Jersey
  - Research Site, Rochester, New York
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Plymouth Meeting, Pennsylvania
  - Research Site, Johnston, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Bartlett, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Walla Walla, Washington
- Canada (5):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Markham, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Waterloo, Ontario

REFERENCES:
- [Background] Bagel J, Tyring S, Rice KC, Collier DH, Kricorian G, Chung J, Iles J, Stolshek BS, Kaliyaperumal A, Papp KA. Open-label study of etanercept treatment in patients with moderate-to-severe plaque psoriasis who lost a satisfactory response to adalimumab. Br J Dermatol. 2017 Aug;177(2):411-418. doi: 10.1111/bjd.15381. Epub 2017 Jul 19. PMID 28196270
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 48 centers in the United States (US) and Canada. Participants were enrolled from 01 February 2012 until 04 November 2014.
Period: Overall Study
Arm/Group | Etanercept 50 mg
Started | 64
Completed | 56
Not Completed | 8
Not completed — Non-compliance | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 4
Not completed — Requirement for Alternative Therapy | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 40
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Black or African American | 4
  Native Hawaiian or other Pacific Islander | 0
  White | 53
  Multiple | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 7
  Not Hispanic/Latino | 57
Psoriasis Area Severity Index (PASI) [Mean (Standard Deviation); unit: units on a scale] — The psoriasis area and severity index (PASI) score incorporates measures of erythema, desquamation, infiltration, and affected body surface area. Involvement and severity of psoriasis was scored by physicians using a scale from 0 to 72, where 0 = no psoriasis and 72 = severe disease.
  units on a scale | 16.81 (6.86)
Percent of Body Surface Area (BSA) Involved in Psoriasis [Mean (Standard Deviation); unit: percentage of BSA] | 20.90 (16.00)
Static Physician Global Assessment (sPGA) of Psoriasis [Number; unit: participants] — A physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The sPGA of psoriasis comprises a 6-point scale ranging from 0 (clear) to 5 (very severe) with increasing severity.
  participants
    0 = Clear | 0
    1 = Almost clear | 0
    2 = Mild | 0
    3 = Moderate | 50
    4 = Severe | 14
    5 = Very severe | 0
Dermatology Life Quality Index (DLQI) [Mean (Standard Deviation); unit: units on a scale] — The DLQI is a skin disease-specific instrument to evaluate health related quality of life ranging from 0 (best possible score) to 30 (worst possible score). Data were available for 63 participants.
  units on a scale | 12.7 (6.7)
Patient Assessment of Flaking [Mean (Standard Deviation); unit: units on a scale] — The severity of psoriasis flaking assessed by the participant on a scale between 0 and 10, with 0 indicating "no flaking at all" and 10 indicating "worst flaking imaginable." Data were available for 63 participants.
  units on a scale | 7.0 (2.3)
Patient Assessment of Itch [Mean (Standard Deviation); unit: units on a scale] — The severity of a participant's itch assessed by the participant on a scale between 0 and 10, with 0 indicating "no itch at all" and 10 indicating "worst itch imaginable." Data were available for 63 participants.
  units on a scale | 6.5 (2.5)
Patient Assessment of Pain [Mean (Standard Deviation); unit: units on a scale] — The severity of the participant's psoriasis pain assessed by the participant on a scale between 0 and 10, with 0 indicating "does not hurt at all" and 10 indicating "worst hurt imaginable." Data were available for 63 participants.
  units on a scale | 5.0 (3.1)
Patient Assessment of Treatment Satisfaction [Number; unit: participants] — Participants indicated their level of satisfaction with the medication's control of psoriasis on a scale from "very dissatisfied" to "very satisfied". The response scale was adapted from the Medical Outcomes Study: Patient Satisfaction Survey.
  participants
    Very dissatisfied | 24
    Dissatisfied | 14
    Neither satisfied nor dissatisfied | 20
    Satisfied | 2
    Very satisfied | 2
    Missing | 2
Anti-adalimumab Antibody Status at Screening [Number; unit: participants]
  Negative | 21
  Positive | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an sPGA Score of 0 (Clear) or 1 (Almost Clear) at Week 12
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). A sPGA response is defined as a sPGA value of clear (score 0) or almost clear (score 1).
Time Frame: Week 12
Population: The primary analysis set (all participants who received at least one dose of investigational product during the study) with at least 1 post-baseline value. Participants with missing post-baseline data were imputed using the last observation carried forward (LOCF) method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
percentage of participants | 39.7 [27.6 to 52.8]

2. Primary Outcome: Percentage of Participants With an sPGA Score of 0 (Clear) or 1 (Almost Clear) at Week 12 by Anti-adalimumab Antibody Status
Description: as for outcome 1
Time Frame: Week 12
Population: The primary analysis set with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Anti-adalimumab Antibody Positive: Participants who were anti-adalimumab antibody positive at screening received etanercept 50 mg, BIW, subcutaneously for 12 weeks followed by 50 mg, QW for an additional 12 weeks.
- Anti-adalimumab Antibody Negative: Participants who were anti-adalimumab antibody negative at screening received etanercept 50 mg, twice weekly (BIW), subcutaneously (SC) for 12 weeks followed by 50 mg, once weekly (QW), SC for an additional 12 weeks.
Arm/Group | Anti-adalimumab Antibody Positive | Anti-adalimumab Antibody Negative
Number analyzed (Participants) | 40 | 20
percentage of participants | 45.0 [29.26 to 61.51] | 35.0 [15.39 to 59.22]
Statistical Analysis 1: Comparison: Anti-adalimumab Antibody Positive vs Anti-adalimumab Antibody Negative; Test type: Superiority or Other; p = 0.4505, Wald asymptotic test; Difference = 10.00, 95% CI 2-sided [-15.97 to 35.97]

3. Secondary Outcome: Percentage of Participants With an sPGA Score of 0 (Clear) or 1 (Almost Clear) at All Other Visits
Description: as for outcome 1
Time Frame: Weeks 4, 8, 16, 20 and 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
percentage of participants
  Week 4 | 4.8 [1.0 to 13.3]
  Week 8 | 23.8 [14.0 to 36.2]
  Week 16 | 39.7 [27.6 to 52.8]
  Week 20 | 42.9 [30.5 to 56.0]
  Week 24 | 38.1 [26.1 to 51.2]

4. Secondary Outcome: Percentage of Participants With an sPGA Score of 0 (Clear) or 1 (Almost Clear) at All Other Visits by Anti-adalimumab Antibody Status
Description: as for outcome 1
Time Frame: Weeks 4, 8, 16, 20 and 24
Population: Primary analysis set participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Anti-adalimumab Antibody Negative: Participants who were anti-adalimumab antibody negative at screening received etanercept 50 mg, BIW, subcutaneously for 12 weeks followed by 50 mg, QW for an additional 12 weeks.
Arm/Group | Anti-adalimumab Antibody Positive | Anti-adalimumab Antibody Negative
Number analyzed (Participants) | 43 | 21
percentage of participants
  Week 4 (n = 42, 21) | 4.8 [0.58 to 16.16] | 4.8 [0.12 to 23.82]
  Week 8 (n = 39, 21) | 17.9 [7.54 to 33.53] | 38.1 [18.11 to 61.56]
  Week 16 (n = 37, 19) | 37.8 [22.46 to 55.24] | 42.1 [20.25 to 66.50]
  Week 20 (n = 38, 19) | 44.7 [28.62 to 61.70] | 47.4 [24.45 to 71.14]
  Week 24 (n = 37, 18) | 40.5 [24.75 to 57.90] | 38.9 [17.30 to 64.25]

5. Secondary Outcome: Percentage of Participants With an sPGA Score of 0, 1 or 2 at Each Visit
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). The percentage of participants with a score of 0 (clear), 1 (almost clear) or 2 (mild) is reported.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
percentage of participants
  Week 4 | 52.4 [39.4 to 65.1]
  Week 8 | 71.4 [58.7 to 82.1]
  Week 12 | 84.1 [72.7 to 92.1]
  Week 16 | 76.2 [63.8 to 86.0]
  Week 20 | 76.2 [63.8 to 86.0]
  Week 24 | 73.0 [60.3 to 83.4]

6. Secondary Outcome: Percentage of Participants With an sPGA Score of 0, 1 or 2 by Anti-adalimumab Antibody Status at Each Visit
Description: as for outcome 5
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anti-adalimumab Antibody Positive | Anti-adalimumab Antibody Negative
Number analyzed (Participants) | 43 | 21
percentage of participants
  Week 4 (n = 42, 21) | 45.2 [29.85 to 61.33] | 66.7 [43.03 to 85.41]
  Week 8 (n = 39, 21) | 61.5 [44.62 to 76.64] | 90.5 [69.62 to 98.83]
  Week 12 (n = 40, 20) | 85.0 [70.16 to 94.29] | 95.0 [75.13 to 99.87]
  Week 16 (n = 37, 19) | 81.1 [64.84 to 92.04] | 73.7 [48.80 to 90.85]
  Week 20 (n = 38, 19) | 81.6 [65.67 to 92.26] | 78.9 [54.43 to 93.95]
  Week 24 (n = 37, 18) | 78.4 [61.79 to 90.17] | 77.8 [52.36 to 93.59]

7. Secondary Outcome: Static Physician Global Assessment (sPGA) at Each Visit
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema).
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
units on a scale
  Week 4 | 2.5 (0.7) [39.4 to 65.1]
  Week 8 | 2.1 (0.8) [58.7 to 82.1]
  Week 12 | 1.7 (0.9) [72.7 to 92.1]
  Week 16 | 1.8 (1.0) [63.8 to 86.0]
  Week 20 | 1.7 (1.0) [63.8 to 86.0]
  Week 24 | 1.8 (1.0) [60.3 to 83.4]

8. Secondary Outcome: Static Physician Global Assessment (sPGA) by Anti-adalimumab Antibody Status at Each Visit
Description: as for outcome 7
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-adalimumab Antibody Positive | Anti-adalimumab Antibody Negative
Number analyzed (Participants) | 43 | 21
units on a scale
  Week 4 (n = 42, 21) | 2.57 (0.11) [39.4 to 65.1] | 2.29 (0.12)
  Week 8 (n = 39, 21) | 2.23 (0.14) [58.7 to 82.1] | 1.71 (0.14)
  Week 12 (n = 40, 20) | 1.68 (0.14) [72.7 to 92.1] | 1.55 (0.18)
  Week 16 (n = 37, 19) | 1.73 (0.14) [63.8 to 86.0] | 1.74 (0.23)
  Week 20 (n = 38, 19) | 1.63 (0.15) [63.8 to 86.0] | 1.63 (0.22)
  Week 24 (n = 37, 18) | 1.73 (0.16) [60.3 to 83.4] | 1.83 (0.23)

9. Secondary Outcome: Percentage of Participants With a PASI 50 Response at Each Visit
Description: A PASI 50 response is a 50% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0 to 72, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
percentage of participants
  Week 4 | 30.2 [19.2 to 43.0]
  Week 8 | 61.9 [48.8 to 73.9]
  Week 12 | 77.8 [65.5 to 87.3]
  Week 16 | 79.4 [67.3 to 88.5]
  Week 20 | 81.0 [69.1 to 89.8]
  Week 24 | 81.0 [69.1 to 89.8]

10. Secondary Outcome: Percentage of Participants With a PASI 50 Response by Anti-adalimumab Antibody Status at Each Visit
Description: as for outcome 9
Time Frame: Baseline and weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anti-adalimumab Antibody Positive | Anti-adalimumab Antibody Negative
Number analyzed (Participants) | 43 | 21
percentage of participants
  Week 4 (n = 42, 21) | 21.4 [10.30 to 36.81] | 47.6 [25.71 to 70.22]
  Week 8 (n = 39, 21) | 59.0 [42.10 to 74.43] | 76.2 [52.83 to 91.78]
  Week 12 (n = 40, 20) | 72.5 [56.11 to 85.40] | 100.0 [83.16 to 100.00]
  Week 16 (n = 37, 19) | 78.4 [61.79 to 90.17] | 89.5 [66.86 to 98.70]
  Week 20 (n = 38, 19) | 84.2 [68.75 to 93.98] | 89.5 [66.86 to 98.70]
  Week 24 (n = 37, 18) | 86.5 [71.23 to 95.46] | 88.9 [65.29 to 98.62]

11. Secondary Outcome: Percentage of Participants With a PASI 75 Response at Each Visit
Description: A PASI 75 response is a 75% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0 to 72, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
percentage of participants
  Week 4 | 4.8 [1.0 to 13.3]
  Week 8 | 25.4 [15.3 to 37.9]
  Week 12 | 46.0 [33.4 to 59.1]
  Week 16 | 49.2 [36.4 to 62.1]
  Week 20 | 50.8 [37.9 to 63.6]
  Week 24 | 47.6 [34.9 to 60.6]

12. Secondary Outcome: Percentage of Participants With a PASI 75 Response by Anti-adalimumab Antibody Status at Each Visit
Description: as for outcome 11
Time Frame: Baseline and weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anti-adalimumab Antibody Positive | Anti-adalimumab Antibody Negative
Number analyzed (Participants) | 43 | 21
percentage of participants
  Week 4 (n = 42, 21) | 2.4 [0.06 to 12.57] | 9.5 [1.17 to 30.38]
  Week 8 (n = 39, 21) | 20.5 [9.30 to 36.46] | 38.1 [18.11 to 61.56]
  Week 12 (n = 40, 20) | 47.5 [31.51 to 63.87] | 50.0 [27.20 to 72.80]
  Week 16 (n = 37, 19) | 51.4 [34.40 to 68.08] | 47.4 [24.45 to 71.14]
  Week 20 (n = 38, 19) | 55.3 [38.30 to 71.38] | 52.6 [28.86 to 75.55]
  Week 24 (n = 37, 18) | 56.8 [39.49 to 72.90] | 38.9 [17.30 to 64.25]

13. Secondary Outcome: Percentage of Participants With a PASI 90 Response at Each Visit
Description: A PASI 90 response is a 90% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0 to 72, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
percentage of participants
  Week 4 | 0 [0.0 to 5.7]
  Week 8 | 3.2 [0.4 to 11.0]
  Week 12 | 22.2 [12.7 to 34.5]
  Week 16 | 25.4 [15.3 to 37.9]
  Week 20 | 19.0 [10.2 to 30.9]
  Week 24 | 23.8 [14.0 to 36.2]

14. Secondary Outcome: Percentage of Participants With a PASI 90 Response by Anti-adalimumab Antibody Status at Each Visit
Description: as for outcome 13
Time Frame: Baseline and weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anti-adalimumab Antibody Positive | Anti-adalimumab Antibody Negative
Number analyzed (Participants) | 43 | 21
percentage of participants
  Week 4 (n = 42, 21) | 0 [0.00 to 8.41] | 0 [0.00 to 16.11]
  Week 8 (n = 39, 21) | 5.1 [0.63 to 17.32] | 0 [0.00 to 16.11]
  Week 12 (n = 40, 20) | 27.5 [14.60 to 43.89] | 15.0 [3.21 to 37.89]
  Week 16 (n = 37, 19) | 27.0 [13.79 to 44.12] | 21.1 [6.05 to 45.57]
  Week 20 (n = 38, 19) | 23.7 [11.44 to 40.24] | 15.8 [3.38 to 39.58]
  Week 24 (n = 37, 18) | 32.4 [18.01 to 49.79] | 11.1 [1.38 to 34.71]

15. Secondary Outcome: Percentage of Participants With at Least a 1 Grade Improvement in sPGA From Baseline
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). The percentage of participants with an improvement from baseline of ≥ 1 grade is reported.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
percentage of participants
  Week 4 | 65.1 [52.0 to 76.7]
  Week 8 | 79.4 [67.3 to 88.5]
  Week 12 | 85.7 [74.6 to 93.3]
  Week 16 | 79.4 [67.3 to 88.5]
  Week 20 | 77.8 [65.5 to 87.3]
  Week 24 | 76.2 [63.8 to 86.0]

16. Secondary Outcome: Percentage of Participants With at Least a 1 Grade Improvement in sPGA From Baseline by Anti-adalimumab Antibody Status
Description: as for outcome 15
Time Frame: Baseline and weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anti-adalimumab Antibody Positive | Anti-adalimumab Antibody Negative
Number analyzed (Participants) | 43 | 21
percentage of participants
  Week 4 (n = 42, 21) | 64.3 [48.03 to 78.45] | 66.7 [43.03 to 85.41]
  Week 8 (n = 39, 21) | 74.4 [57.87 to 86.96] | 90.5 [69.62 to 98.83]
  Week 12 (n = 40, 20) | 87.5 [73.20 to 95.81] | 95.0 [75.13 to 99.87]
  Week 16 (n = 37, 19) | 86.5 [71.23 to 95.46] | 73.7 [48.80 to 90.85]
  Week 20 (n = 38, 19) | 84.2 [68.75 to 93.98] | 78.9 [54.43 to 93.95]
  Week 24 (n = 37, 18) | 83.8 [67.99 to 93.81] | 77.8 [52.36 to 93.59]

17. Secondary Outcome: Percentage of Participants With at Least a 2 Grade Improvement in sPGA From Baseline
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). The percentage of participants with an improvement from baseline of ≥ 2 grades is reported.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
percentage of participants
  Week 4 | 9.5 [3.6 to 19.6]
  Week 8 | 31.7 [20.6 to 44.7]
  Week 12 | 54.0 [40.9 to 66.6]
  Week 16 | 52.4 [39.4 to 65.1]
  Week 20 | 52.4 [39.4 to 65.1]
  Week 24 | 49.2 [36.4 to 62.1]

18. Secondary Outcome: Percentage of Participants With at Least a 2 Grade Improvement in sPGA From Baseline by Anti-adalimumab Antibody Status
Description: as for outcome 17
Time Frame: Baseline and weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anti-adalimumab Antibody Positive | Anti-adalimumab Antibody Negative
Number analyzed (Participants) | 43 | 21
percentage of participants
  Week 4 (n = 42, 21) | 11.9 [3.98 to 25.63] | 4.8 [0.12 to 23.82]
  Week 8 (n = 39, 21) | 30.8 [17.02 to 47.57] | 38.1 [18.11 to 61.56]
  Week 12 (n = 40, 20) | 67.5 [50.87 to 81.43] | 35.0 [15.39 to 59.22]
  Week 16 (n = 37, 19) | 59.5 [42.10 to 75.25] | 42.1 [20.25 to 66.50]
  Week 20 (n = 38, 19) | 60.5 [43.39 to 75.96] | 47.4 [24.45 to 71.14]
  Week 24 (n = 37, 18) | 59.5 [42.10 to 75.25] | 38.9 [17.30 to 64.25]

19. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI)
Description: The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0 to 72, with higher scores indicating greater severity and/or more extensive psoriasis. Percent change from baseline was calculated as (Baseline Value - Post-baseline Value) / Baseline Value * 100, hence a positive value indicates improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
percent change
  Week 4 | 36.02 (22.09) [19.2 to 43.0]
  Week 8 | 55.33 (25.25) [48.8 to 73.9]
  Week 12 | 67.97 (24.20) [65.5 to 87.3]
  Week 16 | 67.98 (29.83) [67.3 to 88.5]
  Week 20 | 69.58 (26.16) [69.1 to 89.8]
  Week 24 | 67.25 (30.41) [69.1 to 89.8]

20. Secondary Outcome: Percent Change From Baseline in PASI by Anti-adalimumab Antibody Status
Description: as for outcome 19
Time Frame: Baseline and weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with available data
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Anti-adalimumab Antibody Positive | Anti-adalimumab Antibody Negative
Number analyzed (Participants) | 43 | 21
percent change
  Week 4 (n = 42, 21) | 33.38 (3.32) [39.4 to 65.1] | 42.29 (4.98)
  Week 8 (n = 39, 21) | 55.90 (3.93) [58.7 to 82.1] | 59.33 (5.33)
  Week 12 (n = 40, 20) | 69.99 (3.49) [72.7 to 92.1] | 73.71 (3.12)
  Week 16 (n = 37, 19) | 70.76 (3.60) [63.8 to 86.0] | 67.31 (8.78)
  Week 20 (n = 38, 19) | 73.47 (3.75) [63.8 to 86.0] | 72.79 (5.22)
  Week 24 (n = 37, 18) | 73.34 (3.57) [60.3 to 83.4] | 65.71 (9.03)

21. Secondary Outcome: Percent Change From Baseline in the Percentage of Body Surface Area (BSA) Involved With Psoriasis
Description: A measurement of psoriasis involvement, given as the physician's assessment of the percentage of the participant's total body surface area (BSA) involved with psoriasis. The percent of BSA affected was estimated by assuming that the participant's palm, excluding the fingers and thumb, represented roughly 1% of the body's surface. Percent change from baseline was calculated as (Baseline Value - Post-baseline Value) / Baseline Value * 100, hence a positive value indicates improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
percent change
  Week 4 | 19.38 (29.43) [19.2 to 43.0]
  Week 8 | 37.86 (32.50) [48.8 to 73.9]
  Week 12 | 53.82 (32.66) [65.5 to 87.3]
  Week 16 | 60.36 (29.48) [67.3 to 88.5]
  Week 20 | 60.33 (29.79) [69.1 to 89.8]
  Week 24 | 58.13 (34.40) [69.1 to 89.8]

22. Secondary Outcome: Percent Change From Baseline in the Percentage of BSA Involved With Psoriasis by Anti-adalimumab Antibody Status
Description: as for outcome 21
Time Frame: Baseline and weeks 4, 8, 12, 16, 20 and 24
Population: Primary analysis set participants with available data
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Anti-adalimumab Antibody Positive | Anti-adalimumab Antibody Negative
Number analyzed (Participants) | 43 | 21
percent change
  Week 4 (n = 42, 21) | 24.41 (3.99) [39.4 to 65.1] | 15.32 (7.83)
  Week 8 (n = 39, 21) | 40.34 (5.32) [58.7 to 82.1] | 34.36 (7.23)
  Week 12 (n = 40, 20) | 58.58 (4.72) [72.7 to 92.1] | 50.91 (8.00)
  Week 16 (n = 37, 19) | 61.21 (4.83) [63.8 to 86.0] | 63.14 (5.19)
  Week 20 (n = 38, 19) | 65.56 (4.75) [63.8 to 86.0] | 60.11 (5.68)
  Week 24 (n = 37, 18) | 65.30 (5.68) [60.3 to 83.4] | 52.72 (6.99)

23. Secondary Outcome: Patient Satisfaction With Treatment at Week 12
Description: Participants indicated their level of satisfaction with the medication's control of psoriasis on a scale from "very dissatisfied" to "very satisfied".
Time Frame: Week 12
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 61
percentage of participants
  Very dissatisfied | 3.3 (0.4) [0.4 to 11.3]
  Dissatisfied | 13.1 (0.8) [5.8 to 24.2]
  Neither satisfied nor dissatisfied | 21.3 (0.9) [11.9 to 33.7]
  Satisfied | 29.5 [18.5 to 42.6]
  Very satisfied | 32.8 [21.3 to 46.0]

24. Secondary Outcome: Patient Satisfaction With Treatment at Week 24
Description: as for outcome 23
Time Frame: Week 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 62
percentage of participants
  Very dissatisfied | 9.7 (0.4) [3.6 to 19.9]
  Dissatisfied | 21.0 (0.8) [11.7 to 33.2]
  Neither satisfied nor dissatisfied | 16.1 (0.9) [8.0 to 27.7]
  Satisfied | 29.0 [18.2 to 41.9]
  Very satisfied | 24.2 [14.2 to 36.7]

25. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score
Description: The dermatology life quality index (DLQI) is a skin disease-specific instrument to evaluate health-related quality of life. The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answered 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is from 0 (best possible score) to 30 (worst possible score). Change from baseline was calculated as Baseline Value - Post-baseline Value, hence a positive change indicates improvement.
Time Frame: Baseline and Weeks 12 and 24
Population: Primary analysis set participants with at least 1 post-baseline value; LOCF imputation was used. n indicates the number of participants included in the analysis at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 61
units on a scale
  Week 12 (n = 60) | 7.9 (7.9)
  Week 24 (n = 61) | 7.0 (7.3)

26. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI)
Description: The impact of disease severity on the participant's ability to participate in work and other activities was evaluated using the WPAI. WPAI consists of six questions to assess whether the participant was currently employed (Q1); how many hours from work were missed due to problems associated with psoriasis (Q2) or any other reason (Q3); hours actually worked (Q4); degree that psoriasis affected productivity while working (Q5); and degree that psoriasis affected regular activities (Q6) over the past 7 days. Four separate overall scores were calculated, including absenteeism (work time missed due to health), presenteeism (impairment at work due to health), work productivity loss (overall work impairment due to health), and activity impairment due to health. Each score ranges from 0 to 100 with higher scores indicating greater impairment and less productivity. Change from baseline was calculated as Baseline Value - Post-baseline Value, hence a positive change indicates improvement.
Time Frame: Baseline and Weeks 12 and 24
Population: Primary analysis set participants with at least 1 post-baseline value and who were employed (for the first 3 scores); LOCF imputation was used. n indicates the number of participants included in the analysis at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
units on a scale
  Week 12: Absenteeism (n = 43) | 1.35 (5.03)
  Week 24: Absenteeism (n = 43) | -1.62 (15.87)
  Week 12: Presenteeism (n = 38) | 14.47 (24.24)
  Week 24: Presenteeism (n = 41) | 11.22 (19.65)
  Week 12: Work Productivity Loss (n = 43) | 13.13 (25.12)
  Week 24: Work Productivity Loss (n = 43) | 8.93 (21.68)
  Week 12: Activity Impairment (n = 60) | 24.17 (29.24)
  Week 24: Activity Impairment (n = 61) | 17.87 (26.59)

27. Secondary Outcome: Change From Baseline in Patient Assessment of Itch
Description: The severity of the participants itch was individually assessed by the participant. Participants were asked to circle a number between 0 and 10 to describe their itch, with 0 indicating "no itch at all" and 10 indicating "worst itch imaginable." Change from baseline was calculated as Baseline Value - Post-baseline Value, hence a positive change indicates improvement.
Time Frame: Baseline and Week 12 and 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
units on a scale
  Week 12 (n = 60) | 3.9 (2.8)
  Week 24 (n = 61) | 3.5 (3.4)

28. Secondary Outcome: Change From Baseline in Patient Assessment of Pain
Description: The severity of the participants pain was individually assessed by the participant. Participants were asked to circle a number between 0 and 10 to describe how much their psoriasis hurts today, with 0 indicating "does not hurt at all" and 10 indicating "worst hurt imaginable." Change from baseline was calculated as Baseline Value - Post-baseline Value, hence a positive change indicates improvement.
Time Frame: Baseline and Week 12 and 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
units on a scale
  Week 12 (n = 60) | 3.4 (3.1)
  Week 24 (n = 61) | 3.0 (3.4)

29. Secondary Outcome: Change From Baseline in Patient Assessment of Flaking
Description: The severity of the participants pain was individually assessed by the participant. Participants were asked to circle a number between 0 and 10 to describe their flaking, with 0 indicating "no flaking at all" and 10 indicating "worst flaking imaginable." Change from baseline was calculated as Baseline Value - Post-baseline Value, hence a positive change indicates improvement.
Time Frame: Baseline and Week 12 and 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 63
units on a scale
  Week 12 (n = 60) | 4.2 (3.2)
  Week 24 (n = 61) | 3.6 (3.6)

30. Secondary Outcome: Number of Participants With Adverse Events
Description: A treatment-related adverse event is defined as an event that is deemed by the investigator to be related to investigational product.
Time Frame: From first dose of study drug until 30 days after the last dose (up to 28 weeks)
Population: Primary analysis set
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg
Number analyzed (Participants) | 64
participants
  Any adverse event (AE) | 40
  Serious adverse events | 2
  AE leading to discontinuation of study drug | 1
  AE leading to discontinuation from study | 1
  Fatal adverse events | 0
  Treatment-related adverse events (TRAE) | 16
  Serious treatment-related adverse events | 1
  TRAE leading to discontinuation of study drug | 1
  TRAE leading to discontinuation from study | 1
  Fatal treatment-related adverse events | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days after the last dose (up to 28 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Etanercept 50mg BIW/50mg QW: Participants received etanercept 50 mg, twice weekly (BIW), subcutaneously (SC) for 12 weeks followed by 50 mg, once weekly (QW), SC for an additional 12 weeks.
Arm/Group | Etanercept 50mg BIW/50mg QW
Serious Adverse Events (participants affected / at risk) | 2/64
Other Adverse Events (participants affected / at risk) | 16/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept 50mg BIW/50mg QW (N=64)
Colitis ischaemic (Gastrointestinal disorders) | 1
Diverticulitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept 50mg BIW/50mg QW (N=64)
Nasopharyngitis (Infections and infestations) | 5
Vitamin D deficiency (Metabolism and nutrition disorders) | 5
Headache (Nervous system disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.